CLINICAL TRIAL: NCT03485300
Title: Prevalence of Sub Optimal Anti Coagulation in Patients With Prosthetic Cardiac Valves
Brief Title: The Prevalence of Sub Optimal Anti Coagulation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Sobhy Gerges, Resident hematologist at internal medicine department, Assiut University
Other Study IDs: Sub optimal anti coagulation
Record Dates: First submitted 2018-03-27; First posted 2018-04-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Poor Drug Response
MeSH Terms: interventions — Kidney Function Tests; Food-Drug Interactions; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with chronic liver or kidney diseases: Patients with chronic liver diseases may affect warfarin therapeutic outcome as liver is the site of metabolism of the drug by cytochrome p 450 enzymes so it decrease warfarin absorption
  Kidney diseases also affect the clearance of the drug these patients will undergo liver function tests and kidney function tests
  Interventions: Diagnostic Test: Liver and kidney function tests for patients with chronic liver or kidney diseases
- Non compliance of the patient: Missed dose of the warfarin or intermittent drug intake may affect drug therapeutic outcome as well as changing time of drug administration during the day
  Interventions: Behavioral: Non compliance of the patient
- Drugs or food interactions: Administration of other drugs beside warfarin may affect its therapeutic outcome either by inhibition or synergism certain food may also interfere with warfarin especially vitamin k and c rich food so patients will be followed up for drug or food interactions
  Interventions: Drug: Drug or food interactions

INTERVENTIONS:
Diagnostic Test: Liver and kidney function tests for patients with chronic liver or kidney diseases — Tests will be done to patients with history suggestive of chronic liver or renal diseases or for patients clinically suspected
  Other Names: SGOT - SGPT - albumin; creatinine - urea
  Groups: Patients with chronic liver or kidney diseases
Behavioral: Non compliance of the patient — I will order all my patients to take the drug at 10 am and assure the daily in taking of the dose and they will be followed up
  Other Names: Asking patient about daily intake of the drug in certain time
  Groups: Non compliance of the patient
Drug: Drug or food interactions — The patient will be in contact with the researcher for any drug added with warfarin in case of other co morbidity conditions and follow up his/her CBC and INR for measuring its effect on warfarin finding out the effect of food on warfarin therapeutic outcome
  Other Names: Checking other drugs may be added with warfarin and dietary habits
  Groups: Drugs or food interactions

SUMMARY:
A study on warfarin administration to show whether noncompliance of the patient will affect our target (INR) during therapy or not beside its drug and dietary interactions.

The study will show the prevalence of sub optimal anti coagulation among patients with prosthetic cardiac valves that will undergo warfarin therapy.

DETAILED DESCRIPTION:
Besides the risk of infective endocarditis, thromboembolism from the foreign body structures of the prosthesis remains a major problem, which can be effectively reduced, but not inhibited by the use of oral anticoagulants in patients with prosthetic cardiac valves.

Warfarin as a vitamin k antagonist is widely used to decrease risk of thromboembolism but need strict monitoring for INR to avoid warfarin failure or hemorrhage.

It acts through inhibiting an enzyme called the vitamin K1 2,3 epoxide reductase complex, subunit1 (VKORC1).

All patients with mechanical heart valves need the oral anticoagulation to keep the INR between 2.5:3.5 according to valve type, position and other comorbid conditions.

However some patients need higher than expected doses of warfarin to get their (INR) into the target therapeutic range.

Resistance to warfarin has been described as the inability to prolong the prothrombin time or raise the international normalized ratio (INR) into the therapeutic range when the drug is given at normally prescribed doses.

Resistance is different than warfarin failure ,which is defined as a new thrombotic event despite a therapeutic prothrombin time and INR .

The causes of warfarin resistance can be either acquired from high consumption of vitamin K or C ,decreased absorption or increased clearance of the drug ,dietary or drug interactions or hereditary by genetic factors that result either in faster metabolism of the drug (a form of pharmacokinetic resistance) or in lower activity of the drug (pharmacodynamic resistance).

ELIGIBILITY:
Inclusion Criteria:

All patients of prosthetic cardiac valves undergo warfarin therapy with sub optimal anti coagulation

Exclusion Criteria:

* Refusal of the patients
* Patients with target INR (2.5-3.5)
* Patients with hypoalbumenimia and chronic liver diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with valvular heart diseases undergoing prosthetic cardiac valves surgeries and on warfarin treatment that will come to outpatients clinics for regular follow up in either Assuit University Hospital or Assuit Police Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of the prevalence of sub optimal anti coagulation in patients with prosthetic cardiac valves | 1 year
  Warfarin therapy is needed in patients with prosthetic cardiac valves to obtain the target INR from 2.5-3.5 .
  If some patients with prosthetic cardiac valves have sub optimal anti coagulation with INR less than 2.5 with maximal doses of warfarin the research will measure their prevalence in all patients with prosthetic cardiac valves on warfarin therapy and their will be questionnaire for some causes of sub optimal anti coagulation in those patients.
  The research will fulfill the following questionnaire :
  Does the patient compliance play a role in warfarin therapeutic outcome? Does changing the time of warfarin administration during the day affect its therapeutic outcome? Does administration of other medication with warfarin including contraception affect its therapeutic outcome? Does dietary habits of certain foods during warfarin administration affect its therapeutic outcome?

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Management of Supratherapeutic International Normalized Ratio without Bleeding after Warfarin Use — http://www.ncbi.nlm.nih.gov/pubmed/28680174